CLINICAL TRIAL: NCT04528615
Title: A Randomized Controlled Trial to Test the Effectiveness of Coping With Cancer in the Kitchen, a Nutrition Education Program From Diagnosis and Beyond
Brief Title: Testing the Effectiveness of Coping With Cancer in the Kitchen
Acronym: CCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19048-01
Record Dates: First submitted 2020-08-17; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Cancer; Nutrition Aspect of Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCK In-Person Sessions (Experimental): This group received the in-person CCK intervention.
  Interventions: Behavioral: CCK In-Person Sessions
- CCK Printed Materials (Active Comparator): This group received select printed CCK materials.
  Interventions: Behavioral: CCK Printed Materials

INTERVENTIONS:
Behavioral: CCK In-Person Sessions — This group attended eight weeks of nutrition education-focused experiential learning.
  Arms: CCK In-Person Sessions
Behavioral: CCK Printed Materials — This group did not attend any in-person sessions and was only provided with select CCK written materials.
  Arms: CCK Printed Materials

SUMMARY:
The study was a two-arm, randomized controlled trial in which cancer survivors were evenly assigned to either receive the 8-week CCK in-person nutrition intervention immediately or to become the control group that received a selection of CCK printed materials. The aim was to test the effectiveness of CCK for implementing a healthy plant-based diet and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Need to have ever been diagnosed with cancer to be eligible
* Need to have not participated in a Living Plate cooking program
* Need to be able to attend at least seven of the eight sessions of the series with mandatory first and last sessions
* Need to have completed active cancer treatment (not including hormonal or other similar agents, e.g., tamoxifen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Knowledge about the role of a plant-based diet in cancer risk reduction | 9 weeks
  Change from baseline in knowledge about role of consuming a predominantly plant-based diet and cancer risk. Participants rated their agreement (1 = Strongly disagree; 5 = Strongly agree) with six custom items developed by the research team, e.g., "I understand the benefits of consuming whole grains versus processed grains". A composite score was calculated as the average of the 6 ratings (range 1-5; Cronbach's alpha=.80).
Knowledge about the role of a plant-based diet in cancer risk reduction | 15 weeks
  Change from baseline in knowledge about role of consuming a predominantly plant-based diet and cancer risk. Participants rated their agreement (1 = Strongly disagree; 5 = Strongly agree) with six custom items developed by the research team, e.g., "I understand the benefits of consuming whole grains versus processed grains". A composite score was calculated as the average of the 6 ratings (range 1-5; Cronbach's alpha=.80).
Confidence preparing a variety of plant-based foods | 9 weeks
  Change from baseline in confidence to prepare a variety of plant-based foods. Participants indicated "How sure are you that you could prepare the foods listed below in a tasty way?" (1 = Very unsure; 5 = Very sure). The 14-item scale included: 4 whole grains; 4 beans, seeds and legumes; 3 green leafy vegetables; and 3 mixed foods, e.g. healthy one-pot meals. A composite score was calculated as the average of the 14 items (range 1-5; Cronbach's alpha=.75).
Confidence preparing a variety of plant-based foods | 15 weeks
  Change from baseline in confidence to prepare a variety of plant-based foods. Participants indicated "How sure are you that you could prepare the foods listed below in a tasty way?" (1 = Very unsure; 5 = Very sure). The 14-item scale included: 4 whole grains; 4 beans, seeds and legumes; 3 green leafy vegetables; and 3 mixed foods, e.g. healthy one-pot meals. A composite score was calculated as the average of the 14 items (range 1-5; Cronbach's alpha=.75).
Skills to practice a plant-based diet | 9 weeks
  Change from baseline in skills to practice a plant-based diet. Participants rated their agreement (1 = Strongly disagree; 5 = Strongly agree) with five custom items developed by the research team, e.g., "I am confident that I can create a kitchen environment that makes it easier to store, prepare, and consume fruits, vegetables, whole grains, and beans."; the average of the five ratings was calculated to create a skills composite score (range 1-5; Cronbach's alpha=.88).
Skills to practice a plant-based diet | 15 weeks
  Change from baseline in skills to practice a plant-based diet. Participants rated their agreement (1 = Strongly disagree; 5 = Strongly agree) with five custom items developed by the research team, e.g., "I am confident that I can create a kitchen environment that makes it easier to store, prepare, and consume fruits, vegetables, whole grains, and beans."; the average of the five ratings was calculated to create a skills composite score (range 1-5; Cronbach's alpha=.88).
Barriers to eating more fruits and vegetables and whole grains | 9 weeks
  Change from baseline in barriers to eating more fruits and vegetables and whole grains. We adapted items from an existing barriers instrument to measure perceived barriers to eating more fruits and vegetables (F&V) (average score of 15 items; Cronbach's alpha = .89) and whole grains (average score of 14 items; Cronbach's alpha = .83). Participants were asked the general question, "Listed below are some common reasons why people don't eat more servings of vegetables and fruits each day. Indicate whether or not this is a reason for you by marking how much you agree or disagree." (1 = Strongly disagree; 5 = Strongly agree). In addition, using the same list of possible reasons (excluding spoil too quickly), participants indicated whether it was a common reason they didn't eat more servings of whole grains. Example reasons included: take too much time to prepare; my family doesn't like them; hard to find a variety of good ones.
Barriers to eating more fruits and vegetables and whole grains | 15 weeks
  Change from baseline in barriers to eating more fruits and vegetables. We adapted items from an existing barriers instrument to measure perceived barriers to eating more fruits and vegetables (F&V) (average score of 15 items; Cronbach's alpha = .89) and whole grains (average score of 14 items; Cronbach's alpha = .83). Participants were asked the general question, "Listed below are some common reasons why people don't eat more servings of vegetables and fruits each day. Indicate whether or not this is a reason for you by marking how much you agree or disagree." (1 = Strongly disagree; 5 = Strongly agree). In addition, using the same list of possible reasons (excluding spoil too quickly), participants indicated whether it was a common reason they didn't eat more servings of whole grains. Example reasons included: take too much time to prepare; my family doesn't like them; hard to find a variety of good ones.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Miller, PhD, Principal Investigator — American Institute for Cancer Research
Locations (1):
- Cancer Support Community Los Angeles, Los Angeles, California, United States

REFERENCES:
- See also: Related Info — http://www.aicr.org